CLINICAL TRIAL: NCT03214380
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro, Both in Combination With Insulin Glargine or Insulin Degludec in Adults With Type 2 Diabetes PRONTO-T2D
Brief Title: A Study of LY900014 Compared to Insulin Lispro in Participants With Type 2 Diabetes
Acronym: PRONTO-T2D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16314; I8B-MC-ITRN (Other: Eli Lilly and Company); 2015-005357-12 (EudraCT Number)
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-08-15

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Glargine; insulin degludec; Metformin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY900014 (Experimental): LY900014 given subcutaneously (SC) with each meal with either 100 U/mL (U-100) basal insulin glargine given SC once or twice daily or U-100 or 200 U/mL (U-200) insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec; Drug: Metformin; Drug: SGLT2 inhibitor
- Insulin Lispro (Humalog) (Active Comparator): Insulin lispro given SC with each meal with either U-100 basal insulin glargine given SC once or twice daily or U-100 or U-200 insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec; Drug: Metformin; Drug: SGLT2 inhibitor
- LY900014 Maximum Extended Enrollment (MEE) (Experimental): LY900014 given subcutaneously (SC) with each meal with either U-100 basal insulin glargine given SC once or twice daily or U-100 or U-200 insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec; Drug: Metformin; Drug: SGLT2 inhibitor
- Insulin Lispro (Humalog) MEE (Active Comparator): Insulin lispro given SC with each meal with either U-100 basal insulin glargine given SC once or twice daily or U-100 or U-200 insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec; Drug: Metformin; Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014; LY900014 Maximum Extended Enrollment (MEE)
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog
  Arms: Insulin Lispro (Humalog); Insulin Lispro (Humalog) MEE
Drug: Insulin Glargine — Administered SC
Drug: Insulin Degludec — Administered SC
Drug: Metformin — Administered orally.
Drug: SGLT2 inhibitor — Administered orally.

SUMMARY:
The purpose of this study is to compare LY900014 to insulin lispro, both in combination with insulin glargine or insulin degludec, in participants with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed (clinically) with T2D, based on the World Health Organization (WHO) classification for at least 1 year prior to screening.
* Have been treated for at least 90 days prior to screening with:

  * Basal insulin (insulin glargine U-100 [Basaglar/Abasaglar or LANTUS] or U-300, insulin detemir, insulin degludec U-100 or U-200, or neutral protamine Hagedorn [NPH] insulin) in combination with at least 1 prandial injection of bolus insulin (insulin lispro U-100 or U-200, insulin aspart, insulin glulisine, or regular insulin) Or
  * Premixed analog or human insulin regimens with any basal and bolus insulin combination injected at least twice daily
* Participants may be treated with up to 3 of the following oral antihyperglycemic medications (OAMs) in accordance with local regulations:

  * Metformin
  * Dipeptidyl peptidase-4 (DPP-4) inhibitor
  * Sodium glucose cotransporter 2 (SGLT2) inhibitor
  * Sulfonylurea
  * Meglitinide
  * Alpha-glucoside inhibitor
* Have an HbA1c value between ≥7.0 and ≤10.0%, according to the central laboratory at the time of screening.
* Have a body mass index (BMI) of ≤45.0 kilograms per meter squared at screening.

Exclusion Criteria:

* Have been diagnosed, at any time, with type 1 diabetes (T1D) or Latent Autoimmune Diabetes in Adults.
* Have hypoglycemia unawareness as judged by the investigator.
* Have had any episode of severe hypoglycemia within the 6 months prior to screening.
* Have had 1 or more episodes of diabetic ketoacidosis or hyperglycemic hyperosmolar state within the 6 months prior to screening.
* Have used thiazolidinediones, Glucagon-Like Peptide 1 (GLP-1) receptor agonist, or pramlintide within 90 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (116):
- United States (31):
  - Valley Research, Fresno, California
  - Diabetes and Endocrine Associates, La Mesa, California
  - First Valley Medical Group, Lancaster, California
  - National Research Institute, Los Angeles, California
  - Care Access Research, Santa Clarita, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - The Center For Diabetes & Endocrine Care, Fort Lauderdale, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - East West Medical Institute, Honolulu, Hawaii
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Northwest Clinical Trials, Boise, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Iderc, P.L.C., West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton O'Neil Diabetes and Endocrinology Center, Kansas City, Kansas
  - Palm Research Center, Las Vegas, Nevada
  - Manhattan Medical Research, New York, New York
  - Aventiv Research, Columbus, Ohio
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Partners in Nephrology & Endocrinology, Pittsburgh, Pennsylvania
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Texas Diabetes and Endocrinology-Austin South, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Private: Dr. Larry Stonesifer, Federal Way, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., CABA, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., CABA, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ciudad Autonoma de Buenos Aire, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Mar del Plata, Buenos Aires
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Oaklands Park, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Fremantle, Western Australia
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Prague
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Bad Mergentheim, Baden-Wurttemberg
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Falkensee, Brandenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pohlheim, Hesse
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Münster, North Rhine-Westphalia
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Mayen, Rhineland-Palatinate
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Saint Ingbert-Oberwürzbach, Saarland
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Magdeburg, Saxony-Anhalt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldenburg in Holstein, Schleswig-Holstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
- India (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad, Gujarat
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ahmedabad, Gujarat
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Bangalore, Karnataka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore, Karnataka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Pune, Maharashtra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune, Maharashtra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai, Maharshtra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur, Rajasthan
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Chennai, Tamil Nadu
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Hyderabad, Telangana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabad, Telangana
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Palmero
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sesto San Giovanni
- Japan (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Naka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Tama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamato
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jalisco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- Puerto Rico (5):
  - Centro de Endocrinologia y Nutricion del Turabo, Caguas
  - Manati Center for Clinical Research Inc, Manatí
  - Ponce School of Medicine CAIMED Center, Ponce
  - Research and Cardiovascular Corp., Ponce
  - GCM Medical Group PSC, San Juan
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kursk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
- Slovakia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice, Slovak Republic
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malacky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nové Mesto nad Váhom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Púchov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rožňava
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si, Gyeonggi-do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ansan-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gangwon-do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yongkang District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Piras de Oliveira C, Dellva MA, Bue-Valleskey J, Chang AM, Liao B. Fasting and postprandial plasma glucose contributions to hemoglobin A1c and time in range in people with diabetes on multiple daily injection insulin therapy: Results from the PRONTO-T1D and PRONTO-T2D clinical trials. J Diabetes Complications. 2024 Jan;38(1):108648. doi: 10.1016/j.jdiacomp.2023.108648. Epub 2023 Nov 16. PMID 38035641
- [Derived] Zhang Q, Chigutsa F, Chang AM. Efficacy and Safety of Ultra-Rapid Lispro in Younger and Older Patients with Type 2 Diabetes: Randomized Double-Blind PRONTO-T2D Study. Diabetes Ther. 2022 Aug;13(8):1547-1557. doi: 10.1007/s13300-022-01290-4. Epub 2022 Jul 4. PMID 35781789
- [Derived] Jinnouchi H, Imori M, Nishiyama H, Imaoka T. Ultra-Rapid Lispro Efficacy and Safety Compared to Humalog(R) in Japanese Patients With Type 2 Diabetes: PRONTO-T2D Subpopulation Analysis. Diabetes Ther. 2020 Sep;11(9):2075-2088. doi: 10.1007/s13300-020-00890-2. Epub 2020 Jul 29. PMID 32728833
- [Derived] Blevins T, Zhang Q, Frias JP, Jinnouchi H, Chang AM; PRONTO-T2D Investigators. Randomized Double-Blind Clinical Trial Comparing Ultra Rapid Lispro With Lispro in a Basal-Bolus Regimen in Patients With Type 2 Diabetes: PRONTO-T2D. Diabetes Care. 2020 Dec;43(12):2991-2998. doi: 10.2337/dc19-2550. Epub 2020 Jul 2. PMID 32616612
- See also: A Study of LY900014 Compared to Insulin Lispro in Participants With Type 2 Diabetes (PRONTO-T2D) — https://www.lillytrialguide.com/en-US/studies/type-2-diabetes/ITRN#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The purpose of the Lead-in Period was to titrate basal insulin prior to randomization. Participants were then randomized to receive Insulin lispro (Humalog) or LY900014 in the Treatment Period (Period 2).
Groups:
- Insulin Lispro (Humalog) Lead-In; Insulin Lispro (Humalog): 100 U/mL Insulin lispro given SC with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
- LY900014; LY900014 (MEE): 100 U/mL LY900014 SC with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
- Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment; Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE): 100 U/mL Insulin lispro (Humalog) SC with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
Period: Lead-in
Arm/Group | Insulin Lispro (Humalog) Lead-In | Insulin Lispro (Humalog) | LY900014 | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment | Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE) | LY900014 (MEE)
Started | 750 | 0 | 0 | 183 | 0 | 0
Received at Least 1 Dose Lead-in Insulin | 750 | 0 | 0 | 183 | 0 | 0
Completed | 673 | 0 | 0 | 164 | 0 | 0
Not Completed | 77 | 0 | 0 | 19 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 1 | 0 | 0
Not completed — Eligibility Criteria | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 7 | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 41 | 0 | 0 | 14 | 0 | 0
Not completed — Family Emergency | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Natural Disaster | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Non Compliance | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Schedule | 2 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Insulin Lispro (Humalog) Lead-In | Insulin Lispro (Humalog) | LY900014 | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment | Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE) | LY900014 (MEE)
Started | 0 (Participants received Insulin Lispro during Lead-in Period.) | 337 (Participants were randomized to either LY900014 or Insulin lispro for Intensive Treatment Period.) | 336 (Participants were randomized to either LY900014 or Insulin lispro for Intensive Treatment Period.) | 0 (Participants received Insulin Lispro during Lead-in Period.) | 82 (Participants were randomized to either LY900014 or Insulin lispro for Intensive Treatment Period.) | 82 (Participants were randomized to either LY900014 or Insulin lispro for Intensive Treatment Period.)
Received at Least 1 Dose of Study Drug | 0 | 337 | 336 | 0 | 82 | 82
Completed | 0 | 319 | 320 | 0 | 73 | 71
Not Completed | 0 | 18 | 16 | 0 | 9 | 11
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 10 | 8 | 0 | 7 | 11
Not completed — Death | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 6 | 3 | 0 | 0 | 0
Not completed — Participant schedule | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Treatment Interruption | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | LY900014 | Insulin Lispro (Humalog) MEE | LY900014 Maximum Extended Enrollment (MEE) | Total
Number analyzed (Participants) | 337 | 336 | 82 | 82 | 837
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.2) | 60.2 (9.4) | 56.6 (9.4) | 57.2 (10.1) | 59.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 152 | 47 | 27 | 388
  Male | 175 | 184 | 35 | 55 | 449
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 0 | 0 | 4
  Asian | 81 | 83 | 70 | 69 | 303
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 16 | 14 | 0 | 0 | 30
  White | 229 | 233 | 12 | 13 | 487
  More than one race | 6 | 5 | 0 | 0 | 11
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 29 | 27 | 0 | 0 | 56
  Puerto Rico | 7 | 7 | 0 | 0 | 14
  Hungary | 13 | 15 | 0 | 0 | 28
  United States | 95 | 92 | 0 | 0 | 187
  Czechia | 20 | 20 | 0 | 0 | 40
  Japan | 46 | 47 | 0 | 0 | 93
  India | 9 | 7 | 40 | 44 | 100
  Russia | 14 | 13 | 11 | 12 | 50
  Spain | 16 | 14 | 0 | 0 | 30
  South Korea | 16 | 16 | 21 | 16 | 69
  Taiwan | 7 | 8 | 9 | 9 | 33
  Italy | 4 | 5 | 0 | 0 | 9
  Mexico | 21 | 22 | 1 | 1 | 45
  Slovakia | 14 | 14 | 0 | 0 | 28
  Australia | 7 | 8 | 0 | 0 | 15
  Germany | 19 | 21 | 0 | 0 | 40
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 7.31 (0.71) | 7.27 (0.68) | 7.53 (0.69) | 7.67 (0.89) | 7.35 (0.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) Efficacy Estimand at Week 26
Description: Change from baseline in HbA1c was performed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least 1 post-baseline HbA1c data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (MEE) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Insulin Lispro (Humalog): Insulin lispro given SC with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
- LY900014: LY900014 given subcutaneously (SC) with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily. Prandial insulin doses were individualized and titrated according to protocol-defined targets.
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 335 | 334
percentage of HbA1c | -0.43 (0.042) | -0.38 (0.042)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Non-Inferiority — Non-inferiority Margin = 0.4 for HbA1c; Least Square Mean Difference (LSMean) = 0.06, 95% CI 2-sided [-0.05 to 0.16]

2. Secondary Outcome: 1-hour Postprandial Glucose (PPG) Excursion During Mixed-Meal Tolerance Test (MMTT) Efficacy Estimand
Description: 1-hour PPG excursion during MMTT uses the analysis of covariance (ANCOVA) model with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum) and treatment as fixed effects and baseline as a covariate. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 1-hour PPG excursion data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 307 | 304
milligrams per deciliter (mg/dL) | 74.9 (3.60) | 63.1 (3.60)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -11.8, 95% CI 2-sided [-18.1 to -5.5]

3. Secondary Outcome: 2-hour PPG Excursion During MMTT Efficacy Estimand
Description: 2-hour PPG excursion during MMTT uses the ANCOVA model with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum) and treatment as fixed effects and baseline as a covariate. The efficacy estimand included participant data when baseline and at least one post-baseline measurement were available prior to permanent discontinuation of study drug.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 2-hour PPG excursion data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 306 | 305
mg/dL | 97.8 (4.50) | 80.4 (4.50)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = -17.4, 95% CI 2-sided [-25.3 to -9.5]

4. Secondary Outcome: Rate of Severe Hypoglycemia
Description: Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within a treatment group *36525. Severe hypoglycemia is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. During these episodes, the participant has an altered mental status and cannot assist in his or her own care, or may be semiconscious or unconscious, or experience com with or without seizures, and may require parenteral therapy.
Time Frame: Baseline through Week 26
Population: All randomized participants with evaluable hypoglycemic data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 337 | 336
Events per 100 participant years | 4.19 | 2.44

5. Secondary Outcome: Rate of Documented Symptomatic Hypoglycemia
Description: Documented symptomatic hypoglycemia is an event during which typical symptoms of hypoglycemia are accompanied by blood glucose (BG) of <54 mg/dL [3.0 millimole per liter (mmol/L)]. The rate of documented symptomatic hypoglycemia was estimated by negative binomial model: number of episodes = treatment with log (treatment exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Week 26
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Events per participant per 30 days/year
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 337 | 336
Events per participant per 30 days/year | 1.34 (0.164) | 2.21 (0.318)

6. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG) at Week 26
Description: Change from baseline in 1,5-AG was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The analysis included data collected prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 1,5-AG data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 334 | 331
milligram per liter (mg/L) | 2.15 (0.234) | 1.99 (0.235)

7. Secondary Outcome: Change From Baseline in 10-Point Self-Monitoring Blood Glucose (SMBG) Values at Week 26
Description: Change from baseline in 10-point SMBG values was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The efficacy estimand included participant data when baseline and at least one post-baseline measurement prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline SMBG data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 276 | 270
mg/dL
  Morning Premeal | -0.8 (2.72) | 1.5 (2.74)
  Morning 1-hour Postmeal: number analyzed (Participants) | 271 | 269
  Morning 1-hour Postmeal | -2.0 (3.44) | -14.1 (3.44)
  Morning 2-hour Postmeal: number analyzed (Participants) | 268 | 268
  Morning 2-hour Postmeal | 0.6 (3.38) | -14.9 (3.38)
  Midday Premeal: number analyzed (Participants) | 273 | 268
  Midday Premeal | 2.4 (2.83) | 4.1 (2.84)
  Midday 1-hour Postmeal: number analyzed (Participants) | 266 | 267
  Midday 1-hour Postmeal | 3.0 (3.48) | -2.0 (3.47)
  Midday 2-hour Postmeal: number analyzed (Participants) | 265 | 268
  Midday 2-hour Postmeal | -2.2 (3.28) | -6.5 (3.27)
  Evening Premeal: number analyzed (Participants) | 271 | 269
  Evening Premeal | 7.0 (3.38) | 10.1 (3.38)
  Evening 1-hour Postmeal: number analyzed (Participants) | 264 | 267
  Evening 1-hour Postmeal | -2.1 (3.24) | -3.0 (3.27)
  Evening 2-hour Postmeal: number analyzed (Participants) | 266 | 266
  Evening 2-hour Postmeal | 0.2 (3.68) | -2.1 (3.73)
  Bedtime: number analyzed (Participants) | 244 | 252
  Bedtime | -3.4 (4.00) | -2.2 (4.02)

8. Secondary Outcome: Change From Baseline in Insulin Dose at Week 26
Description: Change from baseline in insulin dose was analyzed using mixed model repeated measures (MMRM) including fixed class effects of treatment, strata (pooled country, type of basal insulin, HbA1c stratum and number of prandial doses at study entry), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline value. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline basal insulin dose data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Units (U)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 330 | 330
Units (U)
  Basal Insulin Dose: number analyzed (Participants) | 317 | 323
  Basal Insulin Dose | 4.2 (0.82) | 4.6 (0.81)
  Prandial Insulin Dose | 8.3 (1.41) | 12.0 (1.41)
  Total Daily Insulin Dose: number analyzed (Participants) | 316 | 321
  Total Daily Insulin Dose | 12.1 (1.93) | 17.3 (1.92)

9. Secondary Outcome: Change From Baseline in Insulin Treatment Satisfaction Questionnaire (ITSQ) Regimen Inconvenience Domain Score at Week 26
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction.
  Change from baseline in ITSQ regimen inconvenience domain score was calculated using the ANCOVA model with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum), and treatment as fixed effects and baseline as covariate. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and post-baseline data. Missing endpoints were imputed by applying the Last Observation Carried Forward (LOCF) method to post-baseline data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 319 | 319
units on a scale | -0.9 (1.36) | -2.4 (1.37)

10. Secondary Outcome: Change From Baseline in ITSQ Lifestyle Flexibility Domain Score at Week 26
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where higher scores indicate better treatment satisfaction.
  Change from baseline in ITSQ lifestyle flexibility domain score was calculated using the ANCOVA model with strata (pooled country, type of basal insulin, number of prandial doses at study entry, and HbA1c stratum), and treatment as fixed effects and baseline as covariate. The analysis included data prior to permanent discontinuation of study drug.
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and post-baseline data. Missing endpoints were imputed by applying the LOCF method to the post-baseline data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Insulin Lispro (Humalog): Insulin lispro given SC with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily.
- LY900014: LY900014 given subcutaneously (SC) with each meal with either basal insulin glargine given SC once or twice daily or insulin degludec given SC once daily.
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 319 | 319
units on a scale | 1.4 (1.60) | 0.2 (1.60)

11. Secondary Outcome: Number of Participants With HbA1c <7%
Description: Number of participants with HbA1c <7% at Week 26.
Time Frame: Week 26
Population: All participants with baseline and one post-baseline observation while on study drug. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 320 | 316
Participants | 168 | 184

ADVERSE EVENTS:
Time Frame: Baseline up to 30 Weeks
Description: All randomized participants.
Arm/Group | Insulin Lispro (Humalog) Lead-In | Insulin Lispro (Humalog) | LY900014 | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment | Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE) | LY900014 (MEE)
All-Cause Mortality (participants affected / at risk) | 0/750 | 1/337 | 2/336 | 0/183 | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 13/750 | 26/337 | 26/336 | 3/183 | 4/82 | 2/82
Other Adverse Events (participants affected / at risk) | 44/750 | 60/337 | 79/336 | 12/183 | 8/82 | 5/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-In (N=750) | Insulin Lispro (Humalog) (N=337) | LY900014 (N=336) | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment (N=183) | Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE) (N=82) | LY900014 (MEE) (N=82)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (6) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric compression (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-In (N=750) | Insulin Lispro (Humalog) (N=337) | LY900014 (N=336) | Insulin Lispro (Humalog) Lead-In Maximum Extended Enrollment (N=183) | Insulin Lispro (Humalog) Maximum Extended Enrollment (MEE) (N=82) | LY900014 (MEE) (N=82)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 10 (10) | 11 (12) | 2 (2) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 23 (25) | 38 (47) | 47 (56) | 7 (7) | 4 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 20 (21) | 27 (29) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03214380/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03214380/SAP_001.pdf